CLINICAL TRIAL: NCT00127517
Title: A Phase II Double Blind, Placebo Controlled, Randomized, > Multicenter Study With AVR118 Solution in Patients With Advanced > Malignancies Who Are Not Candidates for Curative Chemotherapy.
Brief Title: Palliative Care Study in Patients With Advanced Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Company shifted focus
Sponsor: Advanced Viral Research Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AVR118 04-002
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Cancer
Keywords: Oncology; Palliative Care; Advanced Cancer; Palliative Cancer Care
MeSH Terms: conditions — Neoplasms

INTERVENTIONS:
Drug: peptide-nucleic acid solution AVR118

SUMMARY:
The purpose of this study is to determine whether patients with advanced cancers who receive AVR118 solution for injection into the skin can achieve improvement in quality of life. Based on a study in patients with AIDS, possible benefits may include improved appetite and strength; weight gain; improved mood; and decreased fatigue. For the first three weeks, some patients receive AVR118, and others receive placebo (an injection expected to have no benefits). After three weeks, all patients will be offered the opportunity to take injections of AVR118.

DETAILED DESCRIPTION:
Advanced cancers are usually debilitating. There are few treatments available for symptoms of advanced cancers like loss of appetite, decreased strength, fatigue, and change in mood. A Phase II, double blind study comparing treatment with AVR118 to placebo, followed by an open label phase treating all patients with AVR118, will enable the Sponsor to gather data on safety and efficacy of AVR118 in this patient population. Patients aged 18-80 with advanced cancers (excluding central nervous system [CNS] cancers) who are not receiving chemotherapy, or who are receiving single agent, third line (or beyond) chemotherapy, may be eligible to participate.

ELIGIBILITY:
Inclusion Criteria:

* · Histologically confirmed malignancy (excluding central nervous
* system malignancy)
* · Not a candidate for, or refuses, curative anti-neoplastic therapy.
* · Between the ages of 18 and 80.
* · Symptoms of advanced cancer (loss of appetite, fatigue, weakness,
* malaise) that are not attributed to anemia, concomitant illnesses, or
* obstruction or loss of organ function.
* · Karnofsky performance status of ³40%, _<_ 80%.
* · Normal cognition, interpreted as a Mini-Mental State Score of at
* least 20.
* · Life expectancy of >4 months.
* · Decrease in weight of at least 5% over the preceding 6 months, with
* no weight gain over the most recent 30 days
* · Pretreatment laboratory data within 7 days of enrollment (if
* screening labs are done within 3 days of Day 1, they need not be
* repeated on Day 1).
* ¨ Hemoglobin >8.5 g/dL on no, or on stable doses (hematocrit stable
* within 1 gram and dose stable for one month) of Epogen or similar
* medication.
* ¨ Absolute neutrophil count (ANC) ³1,500/mm^3 .
* ¨ Platelets ³50,000/mm^3 .
* ¨ Total bilirubin £1.5 the upper limit of normal (ULN).
* ¨ ALT and AST £2.5 times the ULN, or, if the patient has liver
* metastases, £5 times the ULN.
* ¨ Creatinine £1.5 mg/dL.
* ¨ Fasting blood sugar -<1.2 x ULN
* ¨ Normal T3, T4, TSH
* · Voluntary written informed consent before performance of any
* study-related procedure that is not part of normal medical care.
* · Ability to self-administer subcutaneous medication, or to have an
* assistant who can administer the study medication according to the
* protocol.
* · Female patient is post-menopausal, surgically sterilized, or willing
* to use acceptable methods of birth control (i.e., a hormonal
* contraceptive, intra-uterine device, diaphragm with spermicide, or
* condom with spermicide, or abstinence) for the duration of the study.
* · Male patient agrees to use an acceptable barrier method for
* contraception during the study.
* · If on an antidepressant, the dose must have been stabilized for at
* least 60 days

Exclusion Criteria:

* · Received immunotherapy, radiation therapy or experimental therapy
* within three weeks.
* · Receiving chemotherapy other than third-line, single agent therapy;
* permitted third-line, single agent dose must be stable for at least
* one month.
* · Diabetes requiring insulin or oral hypoglycemic agents.
* · Mechanical reason to be unable to eat, or is reasonably expected to
* develop an obstruction during the next eight weeks
* · Myocardial infarction within six months of enrollment.
* · Uncontrolled brain metastases or central nervous system disease.
* · Major surgery within four weeks of enrollment.
* · Severe allergies to milk or milk products.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2005-03; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Medical Center of Vincennes, Vincennes, Indiana
  - Queens Medical Associates, Fresh Meadows, New York
  - Jacobi Medical Center, The Bronx, New York